CLINICAL TRIAL: NCT04363619
Title: Insights From the Retina on Cerebral Microvascular Dysfunction in Haemorrhagic Stroke. A Prospective Observational Study
Brief Title: Insights From the Retina on Cerebral Microvascular Dysfunction in Haemorrhagic Stroke
Acronym: RETINA-ICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Emanuela Keller, Prof. Dr., University of Zurich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-01524
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Controls (Placebo Comparator)
  Interventions: Diagnostic Test: OCT and OCTA
- ICH (Experimental)
  Interventions: Diagnostic Test: OCT and OCTA
- aSAH (Experimental)
  Interventions: Diagnostic Test: OCT and OCTA

INTERVENTIONS:
Diagnostic Test: OCT and OCTA — Fundoscopy, OCT and OCTA will be performed 4 times in patients

SUMMARY:
Fundoscopy, optical coherence tomography (OCT) and OCT-angiography (OCTA) are established examinations and bear minimal risks. The recognition of retinal microvascular signs will enhance the pathophysiological understanding of the vasculopathy in patients with intracerebral haemorrhage (ICH) and aneurysmatic subarachnoid hemorrhage (aSAH) and might serve as prognostic and diagnostic indicators.

DETAILED DESCRIPTION:
The purpose of the study is to

* To evaluate the feasibility of fundoscopy, OCT and OCTA imaging in the environment of a Neurocritical Care Unit (NCCU)
* To detect, quantify and associate microvascular changes in the retina with signs of micro-vessel disease in ICH and DCI in aSAH

ELIGIBILITY:
Inclusion Criteria:

* All groups

  * Primary ICH or aSAH with symptoms onset < 3 days
  * 18 to unlimited years of age
  * Signed informed consent obtained from legal representative or patient ICH group
  * Primary ICH localized either in basal ganglia, thalamus, pons or cerebellum aSAH group
  * Ruptured aneurysm visualized in contrast-enhanced computed tomography (angio-CT), MRI or cerebral angiography Control group
  * Stroke due to perimesencepahlic subarachnoid hemorrhage, arteriovenous malformation or isolated traumatic brain injury

Exclusion Criteria:

* All groups

  * Cerebral amyloid angiopathy or other neurodegenerative disease
  * History of migraine with aura or ischemic stroke
  * Contraindication for pupil dilation (intracranial hypertension, allergy against mydriatics, angle closure glaucoma)
  * Any pre-existing or manifest ocular condition affecting either the integrity of retinal vessels, transparency of optical media or the risk of acute angle closure glaucoma
  * Concomitant instable critical illness (e.g. sepsis, multi-organ failure)
  * Intracranial pressure > 20mmHg and refractory to cerebrospinal fluid drainage
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
i. Number of fundus photography, OCT, and OCTA examinations with usable and quantifiable results. | From hospital entry up to 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No